CLINICAL TRIAL: NCT01242007
Title: Lung Function Impairment and Postural Spirometry Changes in Ambulatory Myotonic Dystrophy Patients
Brief Title: Postural Spirometry Changes in Ambulatory Myotonic Dystrophy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nancy (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Chenuel /Pr, University of Nancy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UNBC-11102010
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Myotonic Dystrophy
Keywords: Myotonic dystrophy; Steinert's disease
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Supine spirometry — In addition to the current upright lung function evaluation we performed a supine spirometry
  Other Names: Supine lung function testing

SUMMARY:
Myotonic dystrophy Type 1 (MD1, Steinert's disease), an autosomal dominant multisystem disease, is of the most common muscular dystrophies in adults, with a European prevalence of 3-15/100 000. The disease course is progressive, associating muscular weakness, wasting and myotonia. Respiratory dysfunction is common, involving a restrictive ventilatory abnormality and alveolar hypoventilation, originating from respiratory muscle weakness. Depending on the degree of impairment of their lung function, the quality of life and the prognosis of MD1 patients may be very variable. However, time course and prevalence of such respiratory function impairment have not been clearly identified. More importantly, factors able to predict poor respiratory outcome have not been defined and therefore early prognosis can not be assessed during the follow-up of these patients. In other neuromuscular disorders, especially Amyotrophic Lateral Sclerosis (ALS), postural spirometry has been recommended to improve the detection of diaphragmatic involvement and some authors have suggested that the supine fall in the forced vital capacity could be used to initiate noninvasive positive pressure ventilation and predicts some respiratory symptoms.

In a sample of ambulatory patients with MD1, our study was designed to prospectively achieve two aims: 1) to assess the respective prevalence of a ventilatory restrictive pattern, respiratory muscle weakness, hypoxemia and hypercapnia and 2) to evaluate whether postural changes in lung volumes contribute to sensitize the diagnosis of respiratory weakness and could be used as a predictor of poor respiratory function, including hypoxemia, hypercapnia and restrictive ventilatory disease.

DETAILED DESCRIPTION:
Materials and Methods :

Subjects:

Adult ambulatory patients (18 years of age and older) with a clinical diagnosis of myotonic dystrophy type I were investigated prospectively as part of routine follow-up, from april 2008 to june 2010. Patients were clinically evaluated in the department of "Internal Medicine" and lung function was assessed in the department of "Pulmonary Function Testing", both from the University Hospital of Nancy. Pulmonary tests were ordered for clinical indications, not part of a study protocol. The supine evaluation was added of the conventional lung function testing. All individual were examined and categorized according to a standardized five-point muscular-impairment rating scale, in which a score of 1 indicates no muscular impairment, 2 minimal signs without distal weakness except for digit flexors, 3 distal weakness without proximal weakness except for elbow extensors, 4 moderate proximal weakness, and 5 severe weakness (MIRS).

Lung and respiratory muscle function:

All pulmonary function tests met or exceeds applicable standards of the European Respiratory Society / American Thoracic Society.

Spirometry was performed in the upright-seated position and in the supine position. Respiratory function data were compared with the predicted normal values obtained by the European Community for Steel and Coal and expressed as percentage of the normal value. The flow/volume curve and lung volumes were respectively assessed by an open-circuit spirometry and plethysmography.

Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) were both measured in the seated position using a standard flanged mouthpiece.MIP was measured from Residual Volume (RV) and MEP was measured from Total Lung Capacity (TLC), both in a standard manner. The manoeuvres were repeated at least three times, or until two identical readings were obtained, and the best value was taken. Respiratory Muscle Strength (RMS) was defined as the mean of MIP and MEP expressed as a percent of the predicted values.

Arterial sampling and blood gas analysis :

Arterial blood gases were drawn at rest from the radial artery of the nondominant arm while the patient was comfortably seated for at least 10 minutes. A sterile, self-filling and disposable pre-heparinized system was used to take 1.5 ml of arterial blood.

Arterial oxygen partial pressure (PaO2) and arterial carbon dioxide partial pressure (PaCO2) were determined within 10 minutes after sampling. Room temperature and barometric pressure were recorded on a daily basis and were used to adjust calibrations and measurements. Quality control of the blood-gas equipment was performed twice a day, using standard solution.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of myotonic dystrophy type 1
* 18 years of age and older
* must be able to perform reproducible ventilatory manoeuvres

Exclusion Criteria:

* required non-invasive ventilation
* non reproducible spirometry results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Evidence of lung function impairment | 1 year on average (annual regular follow-up)
  Evidence of ventilatory restriction assessed by lung function testing or hypoxemia or hypercapnia assessed by arterial blood gases analysis

SECONDARY OUTCOMES:
predictive factors of lung function impairment | 1 year on average (annual regular follow-up)
  Using results of upright and supine spirometry we intend to define variables that could predict poor respiratory outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Chenuel, MD, PhD, Principal Investigator — University of Nancy
Locations (1):
- University Hospital of Nancy, Vandœuvre-lès-Nancy, France